CLINICAL TRIAL: NCT01751152
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Assess Clinical Efficacy and Safety of NNC0114-0006 in Subjects With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8828-4004; 2012-002432-93 (EudraCT Number); U1111-1130-8441 (Other: WHO)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Inflammation; Crohn's Disease
MeSH Terms: conditions — Inflammation; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0114-0006 (Experimental)
  Interventions: Drug: NNC0114-0006
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0006 — A single i.v. (intravenous, into the vein) dose. At week 12 the possibility to administer an additional open-label dose of NNC0114-0006 will be provided to all subjects irrespective of initial treatment allocation as long as they are not in need of rescue medication, as judged by the clinical investigator.
  Arms: NNC0114-0006
Drug: placebo — A single i.v. (intravenous, into the vein) dose. At week 12 the possibility to administer an additional open-label dose of NNC0114-0006 will be provided to all subjects irrespective of initial treatment allocation as long as they are not in need of rescue medication, as judged by the clinical investigator.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of the trial is to assess clinical efficacy and safety of NNC0114-0006 in subjects with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severely active Crohn's disease, defined as a Crohn's disease activity index (CDAI) of 220-450 (both inclusive) at Visit 2 (Day 0, Dosing), with evidence of inflammation confirmed by a C-reactive protein (CRP) above or equal to 10 mg/L or endoscopic verification (according to endoscopy imaging manual) performed at Visit 1 (Day -28 to -7, Screening)
* Biologic-naïve subjects or biologic-experienced for the treatment of Crohn's disease. Biologic-experienced subjects are eligible if they have not failed more than one marketed biologic therapy for the treatment of Crohn's disease due to lack of efficacy (primary or secondary efficacy failures)

Exclusion Criteria:

* Body mass index (BMI) equal to or above 38.0 kg/m^2
* Any of the following: symptomatic bowel obstruction, short bowel syndrome, ileostomy or colostomy, surgical bowel resection within 6 months prior to randomisation, total colectomy or subtotal colectomy with less than 20 cm colon remaining, any abscesses not adequately treated
* History of dysplasia in the colon
* Any active or ongoing bacterial infections within 4 weeks prior to randomisation, unless treated and resolved with appropriate therapy
* Any history of serious recurrent infections requiring hospitalisation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Crohn's disease activity index (CDAI) | Week 0, week 4

SECONDARY OUTCOMES:
Change in CDAI | Week 0, week 12
Clinical remission, defined as CDAI of less than 150 | At week 8
Change in the inflammatory bowel disease questionnaire (IBDQ) score | Week 0, week 4
Changes in the Short Form Health Survey (SF-36v2) physical and mental component scores | Week 0, week 4
Incidence of adverse events (AEs) | Up to weeks 24 or 36
Incidence of anti-NNC0114-0006 antibodies | Up to weeks 24 or 36

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (23):
- United States (8):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Laguna Hills, California
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Jackson, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
- Bulgaria (2):
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Czechia (3):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Prague
- Poland (2):
  - Novo Nordisk Investigational Site, Częstochowa
  - Novo Nordisk Investigational Site, Szczecin
- Slovakia (3):
  - Novo Nordisk Investigational Site, Banská Bystrica
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Ružomberok
- Spain (5):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com